CLINICAL TRIAL: NCT02355405
Title: Diagnostic Performance of Lung Ultrasound for Perioperative Atelectasis in Adult Patients Undergoing General Anesthesia
Brief Title: Diagnostic Values of Lung Ultrasound for Perioperative Atelectasis
Status: Completed | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: XY3-LUS-8711
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Postoperative Pulmonary Atelectasis
Keywords: lung ultrasound; atelectasis; thoracic computed Tomography
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: lung ultrasound — lung ultrasound investigations were performed right before and after the surgical procedure.
Radiation: thoracic computed tomography — thoracic CT were performed within one hour after the LUS investigation

SUMMARY:
Lung ultrasound offers a novel, reliable and radiation-free tool for diagnosing perioperative atelectasis and evaluating its severity in adult patients undergoing general anesthesia in the operating room.

DETAILED DESCRIPTION:
Atelectases occur in up to 90% of patients undergoing general anesthesia and intubation. The aim of the present observational study was designed to further to evaluate the diagnostic performance of lung ultrasound (LUS) in detection of postoperative atelectasis in adult patients undergoing general anesthesia. Results of LUS as the experimental method will be compared to the results of computed tomography (CT) as the reference technique for the detection of atelectasis. The investigators want to confirm former findings of the appearance of perioperative atelectases and to prove that ultrasound is a valid tool for detection of atelectases.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and older;
2. American Society of Anesthesiologists (ASA) physical status within class I-III;
3. Scheduled for selective neurosurgical operation with general anesthesia;
4. Need of mechanical ventilation more than 2 hours;

Exclusion Criteria:

1. Patients decline to participate;
2. Pregnancy;
3. Previous thoracic procedures (thoracic drain, thoracotomy, thoracoscopy);
4. A history of pulmonary diseases within last two weeks with abnormal manifestation of lung CT (pulmonary parenchyma or/and interstitial lesions );
5. Pneumothorax or subcutaneous emphysema during peri-operation;
6. Patients with a body mass index (BMI) more than 30 kg/m2;
7. Emergency operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing selective neurosurgical operation in Xiangya Hospital or The Third Xiangya Hospital of Central South University
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Correlation between manifestations of atelectasis in lung ultrasound and in thoracic computed tomography. | From 5 minutes before induction of anesthesia to 1 hour after the surgery
  Measurements of lung ultrasound are performed before induction of anesthesia and immediately after finishing the surgery. Lung CTs are performed the day before surgery and within 1 hour after surgery. Outcome measure: comparison of atelectases by lung ultrasound (experimental method) versus by computed tomography (standard method)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan